CLINICAL TRIAL: NCT05673434
Title: A Clinical Study on the Safety and Efficacy of CAR-T Therapy for the TM4SF1-positive Tumors of Digestive System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Ultra-T Immune Therapeutics Co. LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-TM4SF1-01
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Digestive Tumor
Keywords: Neoplasms
MeSH Terms: conditions — Digestive System Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: TM4SF1 positive CAR-T cells for digestive tumors (Experimental): The present study is proposed to study advanced malignant digestive tumors in adults, and the four escalating doses, namely, 0.5~1.0.,1.0~2.0,2.0~3.0 and 3.0~10.0 (×10 ^6/kg), will be given.
  Intervention: Biological: TM4SF1-positive chimeric antigen receptor T-cell therapy
  Interventions: Biological: TM4SF1-positive chimeric antigen receptor T-cell therapy

INTERVENTIONS:
Biological: TM4SF1-positive chimeric antigen receptor T-cell therapy — Specification: 50mL/bag. Storage: The prepared CAR T-cells are cryopreserved in a preserving medium . This product is manufactured under the current good manufacture practices (cGMP) conditions, with restrictions on chemical components, free from animal- or human-derived components and confirming to the United States Pharmacopeia (USP)<71> and <85> regulations.
  Preservation: The frozen CAR T-cells are preserved in the liquid nitrogen transfer tank.
  Usage: The frozen CAR T-cells are preserved at low temperature and transferred to the bedside. The cells are thawed by 36 degrees centigrade to 38 degrees centigrade. water bath. The frozen cells are gently massaged until complete thawing. Then they are transfused back to the patients intravenously. The transfusion will be finished within 10-20 min.

SUMMARY:
Transmembrane 4 L Six Family Member 1 (TM4SF1) is highly expressed in many tumors of digestive system .

The Chimeric Antigen Receptor T-cells (CAR-T) that target TM4SF1 has been generated in our good manufacturing practices (GMP) facility and the anti-tumor effects have been demonstrated in multiple in vitro and in vivo studies.

Clinical studies are proposed here to evaluate the anti-tumor activity of these cell therapy products for treatment of patients with TM4SF1 positive tumors of digestive system. In this study, the safety, tolerance, and preliminary efficacy of CART-TM4SF1 cells will be examined in patients with refractory/recurrent advanced pancreatic cancer, colorectal cancer, gastric cancer or liver cancer.

Clinical and immunological responses will be evaluated about 30 days and last up to 2 years after CAR-T cell infusion.

DETAILED DESCRIPTION:
Background:

While great progress has been made in CAR T-cell therapy for the treatment of hematologic malignancies, its use in solid tumors is still at the exploratory stage.Transmembrane 4 L Six Family Member 1 (TM4SF1) protein mediates signal transduction events that play a role in the regulation of cell development, activation, growth and motility. It is a cell surface antigen and is highly expressed in different carcinomas.The investigators have developed novel TM4SF1-targeting CAR T-cells (CART-TM4SF1 cells) for the treatment of digestive system tumors.

These engineered T-cells can target and kill the TM4SF1-positive tumor cells in vitro or in mice. Both of the CAR molecules contain a safety switch based on epidermal growth factor receptor (EGFR) to ensure the safety.The investigators propose to investigate the feasibility, safety, and efficacy of CART-TM4SF1 cells for digestive system tumors in patients.

Objectives:

Primary objectives:

1. To determine the safety/tolerance dosages and adverse effects of CART-TM4SF1 cells cells in the treatment of TM4SF1-positive recurrent/refractory advanced tumors of digestive system.
2. To preliminarily evaluate the efficacy of CART-TM4SF1 cells in the treatment of TM4SF1-positive recurrent/refractory advanced tumors of digestive system.

Secondary objectives:

1. To determine the pharmacokinetic (PK)/pharmacodynamic (PD) characteristics of CART-TM4SF1 cells in humans.
2. To evaluate the overall survival (OS) and tumor regression after treatment.
3. To assess the life quality of patients

Study population:

The study population includes 12-24 patients with refractory/recurrent advanced digestive system tumors with positive expression of TM4SF1. The subjects will receive four incremental doses (3-6 subjects in each dose group), as well as safety and preliminary efficacy evaluation.

Design:

* This is a single-center open-label clinical study.
* Recruit patients with refractory/recurrent digestive system tumors, with written consent for this study. Perform biopsy to determine the expression of TM4SF1 of the tumor with immuno-histochemistry (IHC).
* Collect peripheral blood mononuclear cell (PBMC) from the patients, isolate and activate the T cells and transfect them with TM4SF1 targeting CAR, expand the transfected T cells as needed, assess the quality and antitumor activity of the CAR-T products in vitro and then transfer them back the patients via systemic or local injections, and follow up closely to collect related results as needed.
* Clinical and immunological responses will be evaluated closely in about 30 days and last up to 2 years after back-transfusion.

ELIGIBILITY:
Inclusion Criteria:

1. The age at the time of signing the informed consent is ≥ 18 years old and ≤ 75 years old, regardless of gender;
2. BMI ≥ 18.5 (weight (kg)/height (m ²）)；
3. The physical condition score of the Eastern Cooperative Oncology Group (ECOG) is ≤ 2 points;
4. The estimated survival time is not less than 12 weeks;
5. Patients confirmed by histology or cytology, who progress after standard treatment failure, or cannot accept/fail patients with advanced solid tumors with standard treatment, such as gastric cancer, colorectal cancer, pancreatic cancer and other digestive system tumors.
6. According to RECIST 1.1 standard, there is at least one measurable lesion, that is, according to CT or MRI cross section on imaging, the long diameter of non lymph node lesions ≥ 10 mm, or the short diameter of lymph node lesions ≥ 15 mm; measurable disease CT scanning of the longest axis of the focus ≥ 10 mm (CT scanning slice thickness ≤ 5 mm), and the measurable part should not be accepted local treatment such as radiotherapy (for lesions located in the previous radiotherapy area, if progress is confirmed, it is also optional target lesion);
7. It has suitable organs and hematopoietic function (It is not allowed to use any blood components, cytokines, leukemic agents, platelet promoting agents and human albumin preparations within 14 days before screening), according to the following laboratory tests:

   1. Color Doppler echocardiography showed normal diastolic function, left ventricular ejection fraction (LVEF) ≥ 50%, and no large amount of pericardial effusion
   2. Finger oxygen saturation>93%；
   3. Neutrophil (ANC) ≥ 1.5 × 10 9 /L；
   4. Platelet count≥75×10 9 /L；
   5. Hemoglobin (HGB)>90g/L；
   6. Absolute lymphocyte count (ALC)≥0.8×10 9 /L；
   7. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal value (ULN) in patients without liver metastasis and ≤ 3.5 times ULN in patients with liver metastasis;
   8. total bilirubin≤1.5 times ULN；
   9. Creatinine ≤ 1.5 times ULN;
   10. Prothrombin time (PT) or international normalized ratio(INR)<1.5 times ULN, and partial thromboplastin time (APTT)<1.5 times ULN.
8. The expression of TM4SF1 is positive, which can be divided into two cases, and it can meet one of the following conditions：

   1. The tumor tissue samples with recurrence at the primary site or presence of the primary site and within 1 year were detected as high expression of TM4SF1 by immunohistochemistry;
   2. The high expression of TM4SF1 was detected by immunohistochemistry after biopsy in non primary tumor metastasis;
9. Women of childbearing age must have negative pregnancy results during screening period and before drenching treatment.
10. The subject voluntarily joined the group and signed the informed consent form, and voluntarily followed the trial treatment scheme and visit plan.

Exclusion Criteria:

1. Subjects with allergic constitution and allergy to immunotherapy or related drugs；
2. Adverse reactions of previous treatment failed to recover to CTCAE v5.0 grade ≤ 1 ；
3. Patients expected to have major surgery during the study period, including the screening period;；
4. Patients with severe autoimmune diseases requiring long-term (more than 2 months) systemic immunosuppressive therapy;；
5. Any unstable systemic disease: including but not limited to unstable angina pectoris, cerebrovascular accident, transient cerebral ischemia (within 6 months before screening), myocardial infarction (within 6 months before screening), congestive heart failure（≥ NYHA Class III）, severe arrhythmia with poor drug control, liver, kidney or metabolic disease, and hypertension beyond control through standard treatment
6. Known or suspected brain metastasis, including central nervous system and spinal cord compression or meningeal metastasis patient；
7. Other active malignant tumors in the past 5 years
8. Patients with active bleeding and thrombotic disease requiring treatment;
9. Patients with pleural and peritoneal effusion who cannot be controlled and need clinical treatment or intervention；
10. Patients who used corticosteroid hormones (prednisone ≥ 20mg/day or other corticosteroid hormones with equivalent dose) and other immunosuppressants with pharmacological dose 7 days before cell collection and 5 days before cell reinfusion in this study；
11. Alcohol dependent persons or those who have a history of drug abuse or drug abuse in the past one year；
12. Subjects with any mental illness that may affect the understanding of informed consent；
13. Patients with acute or chronic active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection; Patients with human immunodeficiency virus (HIV) antibody positive; Patients with treponema pallidum antibody test positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety assessed by Incidence of Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | 2 years
  After CAR-T cell infusion,the investigators will observe the potential adverse events related to the CAR-T cells infusion such as high fever, kidney failure and so on.
  Adverse events are coded according to MedDRA 22.0. List total number of AEs and SAEs; Number of subjects with different types of AEs and SAEs, case-times and incidence.AEs and SAEs are graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTC AE version 5.0).

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
  The ORR is defined as the percentage of participants who achieve partial response (PR) or better according to Response Evaluation Criteria In Solid Tumors（RECIST) criteria.
CAR-T cell testing | 2 years
  The level of CAR-T cells will be tested regularly by Real-time Quantitative Polymerase Chain Reaction Detecting System(qPCR) or Flow cytometry to evaluate the proliferation in vivo and long-term survival

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Park JW, Chen M, Colombo M, Roberts LR, Schwartz M, Chen PJ, Kudo M, Johnson P, Wagner S, Orsini LS, Sherman M. Global patterns of hepatocellular carcinoma management from diagnosis to death: the BRIDGE Study. Liver Int. 2015 Sep;35(9):2155-66. doi: 10.1111/liv.12818. Epub 2015 Mar 25. PMID 25752327
- [Background] Sher YP, Lin SI, Chai KM, Chen IH, Liu SJ. Endoplasmic reticulum-targeting sequence enhanced the cellular immunity of a tumor-associated antigen L6-based DNA vaccine. Am J Cancer Res. 2019 Sep 1;9(9):2028-2036. eCollection 2019. PMID 31598403
- [Background] Gao C, Yao H, Liu H, Feng Y, Yang Z. TM4SF1 is a potential target for anti-invasion and metastasis in ovarian cancer. BMC Cancer. 2019 Mar 15;19(1):237. doi: 10.1186/s12885-019-5417-7. PMID 30876464
- [Background] Gao H, Chakraborty G, Zhang Z, Akalay I, Gadiya M, Gao Y, Sinha S, Hu J, Jiang C, Akram M, Brogi E, Leitinger B, Giancotti FG. Multi-organ Site Metastatic Reactivation Mediated by Non-canonical Discoidin Domain Receptor 1 Signaling. Cell. 2016 Jun 30;166(1):47-62. doi: 10.1016/j.cell.2016.06.009. PMID 27368100
- [Background] Martinez-Romero J, Bueno-Fortes S, Martin-Merino M, Ramirez de Molina A, De Las Rivas J. Survival marker genes of colorectal cancer derived from consistent transcriptomic profiling. BMC Genomics. 2018 Dec 11;19(Suppl 8):857. doi: 10.1186/s12864-018-5193-9. PMID 30537927
- [Background] Park YR, Kim SL, Lee MR, Seo SY, Lee JH, Kim SH, Kim IH, Lee SO, Lee ST, Kim SW. MicroRNA-30a-5p (miR-30a) regulates cell motility and EMT by directly targeting oncogenic TM4SF1 in colorectal cancer. J Cancer Res Clin Oncol. 2017 Oct;143(10):1915-1927. doi: 10.1007/s00432-017-2440-4. Epub 2017 May 20. PMID 28528497
- [Background] Ma YS, Yu F, Zhong XM, Lu GX, Cong XL, Xue SB, Xie WT, Hou LK, Pang LJ, Wu W, Zhang W, Cong LL, Liu T, Long HD, Sun R, Sun HY, Lv ZW, Wu CY, Fu D. miR-30 Family Reduction Maintains Self-Renewal and Promotes Tumorigenesis in NSCLC-Initiating Cells by Targeting Oncogene TM4SF1. Mol Ther. 2018 Dec 5;26(12):2751-2765. doi: 10.1016/j.ymthe.2018.09.006. Epub 2018 Sep 13. PMID 30301667
- [Background] Xue L, Yu X, Jiang X, Deng X, Mao L, Guo L, Fan J, Fan Q, Wang L, Lu SH. TM4SF1 promotes the self-renewal of esophageal cancer stem-like cells and is regulated by miR-141. Oncotarget. 2017 Mar 21;8(12):19274-19284. doi: 10.18632/oncotarget.13866. PMID 27974706
- [Background] Goodman GE, Hellstrom I, Yelton DE, Murray JL, O'Hara S, Meaker E, Zeigler L, Palazollo P, Nicaise C, Usakewicz J, et al. Phase I trial of chimeric (human-mouse) monoclonal antibody L6 in patients with non-small-cell lung, colon, and breast cancer. Cancer Immunol Immunother. 1993;36(4):267-73. doi: 10.1007/BF01740909. PMID 8382560
- [Background] Ziegler LD, Palazzolo P, Cunningham J, Janus M, Itoh K, Hayakawa K, Hellstrom I, Hellstrom KE, Nicaise C, Dennin R, et al. Phase I trial of murine monoclonal antibody L6 in combination with subcutaneous interleukin-2 in patients with advanced carcinoma of the breast, colorectum, and lung. J Clin Oncol. 1992 Sep;10(9):1470-8. doi: 10.1200/JCO.1992.10.9.1470. PMID 1517790
- [Background] Goodman GE, Hellstrom I, Brodzinsky L, Nicaise C, Kulander B, Hummel D, Hellstrom KE. Phase I trial of murine monoclonal antibody L6 in breast, colon, ovarian, and lung cancer. J Clin Oncol. 1990 Jun;8(6):1083-92. doi: 10.1200/JCO.1990.8.6.1083. PMID 2161448
- [Background] Denardo SJ, O'Grady LF, Richman CM, Goldstein DS, O'Donnell RT, Denardo DA, Kroger LA, Lamborn KR, Hellstrom KE, Hellstrom I, Denardo GL. Radioimmunotherapy for advanced breast cancer using I-131-ChL6 antibody. Anticancer Res. 1997 May-Jun;17(3B):1745-51. PMID 9179228
- [Background] Katz SC, Burga RA, McCormack E, Wang LJ, Mooring W, Point GR, Khare PD, Thorn M, Ma Q, Stainken BF, Assanah EO, Davies R, Espat NJ, Junghans RP. Phase I Hepatic Immunotherapy for Metastases Study of Intra-Arterial Chimeric Antigen Receptor-Modified T-cell Therapy for CEA+ Liver Metastases. Clin Cancer Res. 2015 Jul 15;21(14):3149-59. doi: 10.1158/1078-0432.CCR-14-1421. Epub 2015 Apr 7. PMID 25850950
- [Background] Saied A, Licata L, Burga RA, Thorn M, McCormack E, Stainken BF, Assanah EO, Khare PD, Davies R, Espat NJ, Junghans RP, Katz SC. Neutrophil:lymphocyte ratios and serum cytokine changes after hepatic artery chimeric antigen receptor-modified T-cell infusions for liver metastases. Cancer Gene Ther. 2014 Nov;21(11):457-62. doi: 10.1038/cgt.2014.50. Epub 2014 Oct 3. PMID 25277132
- [Background] Ahmed N, Brawley VS, Hegde M, Robertson C, Ghazi A, Gerken C, Liu E, Dakhova O, Ashoori A, Corder A, Gray T, Wu MF, Liu H, Hicks J, Rainusso N, Dotti G, Mei Z, Grilley B, Gee A, Rooney CM, Brenner MK, Heslop HE, Wels WS, Wang LL, Anderson P, Gottschalk S. Human Epidermal Growth Factor Receptor 2 (HER2) -Specific Chimeric Antigen Receptor-Modified T Cells for the Immunotherapy of HER2-Positive Sarcoma. J Clin Oncol. 2015 May 20;33(15):1688-96. doi: 10.1200/JCO.2014.58.0225. Epub 2015 Mar 23. PMID 25800760